CLINICAL TRIAL: NCT01973335
Title: Diamox/Aldactone to Increase the URinary Excretion of Sodium: an Investigational Study in Congestive Heart Failure
Brief Title: Acetazolamide and Spironolactone to Increase Natriuresis in Congestive Heart Failure
Acronym: DIURESIS-CHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Wilfried Mullens, MD PhD, Prof. Dr., Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ZOL-DIURESIS-CHF
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
Keywords: acetazolamide; bumetanide; cardio-renal syndrome; diuretics; heart failure; natriuresis; spironolactone
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — Combined Modality Therapy; Acetazolamide; Sodium Potassium Chloride Symporter Inhibitors; Bumetanide; Spironolactone

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Acetazolamide/low-dose loop diuretics, upfront spironolactone (Experimental): 2x2 factorial design: This group is the experimental group for both study interventions (acetazolamide and upfront spironolactone).
  See interventions for more details.
  Interventions: Drug: Combination therapy with acetazolamide and low-dose loop diuretics; Drug: Upfront therapy with oral spironolactone
- High-dose loop diuretics, upfront spironolactone (Experimental): 2x2 factorial design: This group is the experimental group for the study intervention with upfront spironolactone. This group receives high-dose loop diuretics as an active comparator to the study intervention with acetazolamide.
  See interventions for more details.
  Interventions: Drug: High-dose loop diuretics; Drug: Upfront therapy with oral spironolactone
- Acetazolamide/low-dose loop diuretics, no spironolactone (Experimental): 2x2 factorial design: This group is the experimental group for the study intervention with acetazolamide. This group receives no intervention with regards to the spironolactone arm.
  See interventions for more details.
  Interventions: Drug: Combination therapy with acetazolamide and low-dose loop diuretics
- High-dose loop diuretics, no spironolactone (Active Comparator): 2x2 factorial design: This group receives high-dose loop diuretics as an active comparator to the study intervention with acetazolamide. This group receives no intervention with regards to the spironolactone arm.
  See interventions for more details.
  Interventions: Drug: High-dose loop diuretics

INTERVENTIONS:
Drug: Combination therapy with acetazolamide and low-dose loop diuretics — * Patients receive 500 mg of intravenous acetazolamide immediately after randomization, with 250 mg intravenous acetazolamide administered on each consecutive day in the morning for as long as the patient is considered volume overloaded by his/her treating cardiologist.
  * Patients receive 2 mg of intravenous bumetanide immediately after randomization, with 1 mg intravenous bumetanide administered on each consecutive day in the morning for as long as the patient is considered volume overloaded by his/her treating cardiologist.
  * If diuresis <1,5 L while the patient is still considered volume overloaded by his/her treating cardiologist, the dose of acetazolamide is maintained at 500 mg and the dose of bumetanide is maintained at 2mg.
  In case of therapy-refractory congestion, treatment is at the discretion of the treating physician, but addition of chlorthalidone 50 mg PO is recommended by the investigators as a first-line option.
  Other Names: Diamox (acetazolamide); Burinex/Bumex (loop diuretics)
  Arms: Acetazolamide/low-dose loop diuretics, no spironolactone; Acetazolamide/low-dose loop diuretics, upfront spironolactone
Drug: High-dose loop diuretics — * Patients receive the double of their daily maintenance dose of oral loop diuretics converted to mg bumetanide as an intravenous bolus after randomization.
  * Patients continue to receive this dose daily on the next 3 days divided between two administrations with at least a 6 h interval for as long as they are considered volume overloaded by the treating cardiologist.
  * If diuresis <1,5 L while the patient is still considered volume overloaded by the treating cardiologist, the dose of bumetanide is doubled.
  In case of therapy-refractory congestion, treatment is at the discretion of the treating physician, but addition of chlorthalidone 50 mg PO is recommended by the investigators as a first-line option.
  Other Names: Burinex/Bumex
  Arms: High-dose loop diuretics, no spironolactone; High-dose loop diuretics, upfront spironolactone
Drug: Upfront therapy with oral spironolactone — Patients randomized to this group receive oral spironolactone (25mg) immediately after randomization and in the morning of each subsequent day unless the serum potassium level is >5 mmol/L.
  Note: Investigators and treating physicians are blinded to treatment allocation for this arm, but no matching placebo is provided, so patients are not.
  Other Names: Aldactone
  Arms: Acetazolamide/low-dose loop diuretics, upfront spironolactone; High-dose loop diuretics, upfront spironolactone

SUMMARY:
This study has two primary objectives:

1. To compare combination therapy with acetazolamide and low-dose loop diuretics versus high-dose loop diuretics (standard of care) in patients with acute decompensated heart failure at high risk for diuretic resistance.
2. To demonstrate the safety and efficacy of upfront therapy with spironolactone in addition to loop diuretic therapy in patients with acute decompensated heart failure at high risk for diuretic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years and able to give informed consent
* Clinical diagnosis of acute decompensated heart failure within the previous 8 h
* At least two clinical signs of congestion (edema, ascites, jugular venous distension, or pulmonary vascular congestion on chest radiography)
* Maintenance therapy with oral loop diuretics at a dose of at least 1 mg bumetanide (1 mg bumetanide = 40 mg furosemide = 20 mg torsemide) for at least 1 month before hospital admission
* NT-proBNP >1000 ng/L
* Left ventricular ejection fraction <50%
* At least one out of three of the following criteria:

  * Serum sodium <136 mmol/L
  * Serum urea/creatinine ratio >50 (comparable to a BUN/creatinine ratio >25)
  * Admission serum creatinine increased with >0.3 mg/dL compared to previous value within 3 months before admission

Exclusion Criteria:

* History of cardiac transplantation and/or ventricular assist device
* Concurrent diagnosis of an acute coronary syndrome defined as typical chest pain and/or electrocardiographic changes in addition to a troponin rise >99th percentile
* Mean arterial blood pressure <65 mmHg, or systolic blood pressure <90 mmHg at the moment of admission
* Use of intravenous inotropes, vasopressors or nitroprusside at any time point during the study
* A baseline estimated glomerular filtration rate <15 mL/min/1.73m² according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula at the moment of inclusion
* Use of renal replacement therapy or ultrafiltration before study inclusion
* Treatment with acetazolamide within the previous month
* Treatment with ≥2 mg bumetanide or an equivalent dose during the index hospitalization before randomization
* Use of diuretics, vasopressin antagonists or mineralocorticoid receptor antagonist not specified by the protocol
* Exposure to nephrotoxic agents (i.e. contrast dye) anticipated within 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Mullens, M.D. Ph.D., Principal Investigator — Ziekenhuis Oost-Limburg; Frederik H. Verbrugge, M.D. Ph.D., Principal Investigator — Ziekenhuis Oost-Limburg
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - University Hospital Leuven, Leuven, Vlaams-Brabant

REFERENCES:
- [Result] Verbrugge FH, Martens P, Ameloot K, Haemels V, Penders J, Dupont M, Tang WHW, Droogne W, Mullens W. Spironolactone to increase natriuresis in congestive heart failure with cardiorenal syndrome. Acta Cardiol. 2019 Apr;74(2):100-107. doi: 10.1080/00015385.2018.1455947. Epub 2018 Mar 27. PMID 29587582
- [Result] Verbrugge FH, Martens P, Ameloot K, Haemels V, Penders J, Dupont M, Tang WHW, Droogne W, Mullens W. Acetazolamide to increase natriuresis in congestive heart failure at high risk for diuretic resistance. Eur J Heart Fail. 2019 Nov;21(11):1415-1422. doi: 10.1002/ejhf.1478. Epub 2019 May 9. PMID 31074184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Dates of the recruitment period: 28/12/2013 till 14/03/2017
  * location: emergency services and outpatient cardiology clinic of 2 tertiary care centers (Ziekenhuis Oost-Limburg, Genk, Belgium & UZ Leuven, Leuven, Belgium)
Pre-assignment Details: None, every patient that was enrolled was immediately randomised and started with the protocol of the study.
Groups:
- Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone: * Patients receive 500 mg of intravenous acetazolamide immediately after randomization, with 250 mg intravenous acetazolamide administered on each consecutive day in the morning for as long as the patient is considered volume overloaded by his/her treating cardiologist.
  * Patients receive 2 mg of intravenous bumetanide immediately after randomization, with 1 mg intravenous bumetanide administered on each consecutive day in the morning for as long as the patient is considered volume overloaded by his/her treating cardiologist.
  * Patients receive open-label oral spironolactone at a dose of 25 mg unless serum potassium levels are >5 mmol/L.
- High-dose Loop Diuretics, Upfront Spironolactone: * Patients receive the double of their daily maintenance dose of oral loop diuretics converted to mg bumetanide as an intravenous bolus after randomization.
  * Patients continue to receive this dose daily on the next 3 days divided between two administrations with at least a 6 h interval for as long as they are considered volume overloaded by the treating cardiologist.
  * Patients receive open-label oral spironolactone at a dose of 25 mg unless serum potassium levels are >5 mmol/L.
- Acetazolamide/Low-dose Loop Diuretics, no Spironolactone: * Patients receive 500 mg of intravenous acetazolamide immediately after randomization, with 250 mg intravenous acetazolamide administered on each consecutive day in the morning for as long as the patient is considered volume overloaded by his/her treating cardiologist.
  * Patients receive 2 mg of intravenous bumetanide immediately after randomization, with 1 mg intravenous bumetanide administered on each consecutive day in the morning for as long as the patient is considered volume overloaded by his/her treating cardiologist.
  * Spironolactone use is prohibited during the first 72 h, but encouraged at discharge.
- High-dose Loop Diuretics, no Spironolactone: * Patients receive the double of their daily maintenance dose of oral loop diuretics converted to mg bumetanide as an intravenous bolus after randomization.
  * Patients continue to receive this dose daily on the next 3 days divided between two administrations with at least a 6 h interval for as long as they are considered volume overloaded by the treating cardiologist.
  * Spironolactone use is prohibited during the first 72 h, but encouraged at discharge.
Period: Overall Study
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
Started | 9 | 7 | 9 | 9
Completed | 9 | 7 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone | Total
Number analyzed (Participants) | 9 | 7 | 9 | 9 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 81 (8) | 75 (7) | 81 (5) | 81 (7) | 80 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 3 | 12
  Male | 7 | 5 | 4 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 9 | 7 | 9 | 9 | 34
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 9 | 7 | 9 | 9 | 34
New York Heart Association functional class [Count of Participants; unit: Participants]
  II | 2 | 0 | 0 | 1 | 3
  III | 5 | 3 | 7 | 4 | 19
  IV | 2 | 4 | 2 | 4 | 12
History of ischemic heart disease [Count of Participants; unit: Participants] | 5 | 6 | 3 | 7 | 21
History of atrial fibrillation [Count of Participants; unit: Participants] | 3 | 4 | 7 | 6 | 20
History of diabetes [Count of Participants; unit: Participants] | 3 | 2 | 2 | 3 | 10
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73m²] | 36 (17) | 32 (9) | 35 (16) | 40 (31) | 36 (20)
Renin-angiotensin blocker therapy [Count of Participants; unit: Participants] | 2 | 4 | 5 | 3 | 14
Beta-blocker therapy [Count of Participants; unit: Participants] | 8 | 7 | 8 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Acetazolamide Arm: Natriuresis 24 h
Description: For the acetazolamide arm of the study, the primary end-point is total natriuresis after 24 h (mmol). To assess this, urine is collected for 24 h after the first administration of diuretics according to the study protocol and natriuresis is calculated as the total amount of diuresis (L) multiplied by the urinary sodium concentration (mmol/L). Subsequently, patients receiving acetazolamide and low-dose loop diuretics (both the groups with and without upfront spironolactone together) are compared to patients not receiving acetazolamide but high-dose loop diuretics instead (both the groups with or without upfront spironolactone together)
Time Frame: 24h
Population: 2 patients not analysed because of errors with 24 h urinary collection
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
Number analyzed (Participants) | 8 | 6 | 9 | 9
mmol | 324 (133) | 300 (165) | 211 (96) | 190 (91)
Statistical Analysis 1: Comparison: Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone vs High-dose Loop Diuretics, Upfront Spironolactone vs Acetazolamide/Low-dose Loop Diuretics, no Spironolactone vs High-dose Loop Diuretics, no Spironolactone; 2x2 factorial design: both acetazolamide groups together are compared with both high-dose loop diuretic groups together; Test type: Superiority; p = 0.515, t-test, 2 sided — Not adjusted for multiple comparisons; Mean Difference (Final Values) = 30, 95% CI 2-sided [-63 to 123]

2. Primary Outcome: Spironolactone Arm: Incidence of Hypo- (Serum Potassium <3.5 mmol/L) or Hyperkalemia (Serum Potassium >5.0 mmol/L)
Description: For the spironolactone arm of the study, the primary end-point is the incidence of either hypo- (serum potassium <3.5 mmol/L) or hyperkalemia (serum potassium >5.0 mmol/L) at any of 3 morning blood samples at consecutive days after randomization. Patients receiving upfront spironolactone (both the group receiving acetazolamide+low dose loop diuretics and the group receiving high-dose loop diuretic therapy) are compared with them receiving no spironolactone (both the group receiving acetazolamide+low dose loop diuretics and the group receiving high-dose loop diuretic therapy).
Time Frame: 72h
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
Number analyzed (Participants) | 9 | 7 | 9 | 9
Participants | 1 | 2 | 5 | 2
Statistical Analysis 1: Comparison: Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone vs High-dose Loop Diuretics, Upfront Spironolactone vs Acetazolamide/Low-dose Loop Diuretics, no Spironolactone vs High-dose Loop Diuretics, no Spironolactone; 2x2 factorial design: analysis according to spironolactone use; Test type: Superiority; p = 0.270, Fisher Exact — Not adjusted for multiple comparisons; Risk Difference (RD) = -0.2

3. Secondary Outcome: NT-proBNP Change After 72 h
Description: Relative NT-proBNP change (%) after 72 h compared to baseline.
Time Frame: 72h
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
Number analyzed (Participants) | 9 | 7 | 9 | 9
percentage change from baseline | -20 (36) | -11 (19) | -3 (40) | -6 (51)

4. Secondary Outcome: Number of Participants With Worsening Renal Function
Description: Worsening renal function is defined as a rise in serum creatine >0.3 mg/dL or a >20% decrease in estimated glomerular filtration rate by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula compared to baseline at any time point before 72 h. Serum creatinine values are assessed at three consecutive mornings after study inclusion.
Time Frame: 72h
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
Number analyzed (Participants) | 9 | 7 | 9 | 9
Participants | 2 | 0 | 3 | 0

5. Secondary Outcome: Persistent Renal Impairment
Description: Persistent renal impairment is defined as a persistently elevated serum creatine >0.3mg/dL or >20% decrease in estimated glomerular filtration rate by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula, above the baseline value of the patient and will be assessed on a scheduled follow-up appointment 4 weeks after hospital discharge.
Time Frame: 4 weeks after hospital discharge
Population: 9 patients died or were too sick for follow-up appointment; 9 refused a venous blood sample at the follow-up appointment (protocol violation)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
Number analyzed (Participants) | 5 | 2 | 5 | 4
Participants | 3 | 1 | 0 | 1

6. Secondary Outcome: Peak Plasma Aldosterone Concentration After 72 h
Description: At three consecutive mornings after study inclusion, blood samples will be taken to assess plasma aldosterone levels. The highest value will constitute the peak plasma aldosterone concentration (ng/L).
Time Frame: 72h
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
Number analyzed (Participants) | 9 | 7 | 9 | 9
ng/L | 196 [127 to 338] | 234 [149 to 334] | 302 [165 to 909] | 204 [153 to 756]

7. Secondary Outcome: Peak Plasma Renin Activity After 72 h
Description: At three consecutive mornings after study inclusion, blood samples will be taken to assess plasma renin activity. The highest value will constitute the peak plasma renin activity (ng/mL/h).
Time Frame: 72h
Measure: Median (Inter-Quartile Range); unit: µg/L/h
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
Number analyzed (Participants) | 9 | 7 | 9 | 9
µg/L/h | 3.8 [0.9 to 6.5] | 5.0 [3.8 to 10.2] | 12.0 [0.8 to 34.3] | 2.5 [0.8 to 28.2]

8. Other Pre Specified Outcome: Natriuresis 48 h
Description: Total natriuresis (mmol) after 48 h.
Time Frame: 48h
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Natriuresis 72 h
Description: Total natriuresis (mmol) after 72 h.
Time Frame: 72h
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Diuresis 24 h
Description: Total amount of urine output (L) after 24 h.
Time Frame: 24h
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Diuresis 48 h
Description: Total amount of urine output (L) after 48 h.
Time Frame: 48h
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Diuresis 72 h
Description: Total amount of urine output (L) after 72 h.
Time Frame: 72h
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Weight Change After 72 h
Description: Body weight change after 72 h compared to admission.
Time Frame: 72h
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Visual Analogue Scale Score for Dyspnea After 24 h
Description: Scale name and construct: Visual analogue scale presented as a line with a movable indicator. Far left of the line indicates no dyspnea at all and far right of the line indicates the worst imaginable dyspnea. The participant can move the indicator to one certain point among the line and the investigator can read at the back a number going from 0 to 100 with 0 indicating no dyspnea and 100 the worst imaginable dyspnea.
Time Frame: 24h
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Visual Analogue Scale Score for Dyspnea After 48 h
Time Frame: 48h
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Visual Analogue Scale Score for Dyspnea After 72 h
Time Frame: 72h
Reporting Status: Not Posted

17. Other Pre Specified Outcome: 4-point Likert Scale for Edema After 24 h
Time Frame: 24h
Reporting Status: Not Posted

18. Other Pre Specified Outcome: 4-point Likert Scale for Edema After 48 h
Time Frame: 48h
Reporting Status: Not Posted

19. Other Pre Specified Outcome: 4-point Likert Scale for Edema After 72 h
Time Frame: 72h
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Incidence of Therapy-refractory Congestion
Description: Need for combinational diuretic therapy with thiazide-type diuretics, bail-out ultrafiltration or renal replacement therapy
Time Frame: 72h
Reporting Status: Not Posted

21. Other Pre Specified Outcome: All-cause Mortality
Time Frame: After 1 year of follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Each patient was contacted by phone after 3 months, 6 months, and 12 months. A qualified study nurse assessed whether the patient died or was hospitalized during the previous 3 months. The electronic medical record was used to assess the reason for hospitalizations.
Arm/Group | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone | High-dose Loop Diuretics, Upfront Spironolactone | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone | High-dose Loop Diuretics, no Spironolactone
All-Cause Mortality (participants affected / at risk) | 6/9 | 5/7 | 5/9 | 5/9
Serious Adverse Events (participants affected / at risk) | 3/9 | 5/7 | 2/9 | 3/9
Other Adverse Events (participants affected / at risk) | 6/9 | 4/7 | 7/9 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone (N=9) | High-dose Loop Diuretics, Upfront Spironolactone (N=7) | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone (N=9) | High-dose Loop Diuretics, no Spironolactone (N=9)
Hospital readmission due to heart failure (Cardiac disorders) | 3 | 5 | 2 | 3
Serious hyperkalemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 — Serum potassium level >6.5 mmol/L during the 72 h treatment interval
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acetazolamide/Low-dose Loop Diuretics, Upfront Spironolactone (N=9) | High-dose Loop Diuretics, Upfront Spironolactone (N=7) | Acetazolamide/Low-dose Loop Diuretics, no Spironolactone (N=9) | High-dose Loop Diuretics, no Spironolactone (N=9)
Metabolic acidosis (Renal and urinary disorders) | 2 | 3 | 2 | 3 — Serum bicarbonate level <22.0 mEq/L during the 72 h treatment interval
Moderate hyperkalemia (Renal and urinary disorders) | 0 | 1 | 2 | 0 — Serum potassium level 5.1-6.5 mmol/L during the 72 h treatment interval
Hypokalemia (Renal and urinary disorders) | 1 | 1 | 3 | 2 — Serum potassium level <3.5 mmol/L during the 72 h treatment interval
Worsening renal function (Renal and urinary disorders) | 2 | 0 | 3 | 0 — Increase of the serum creatinine level >0.3 mg/dL during the 72 h treatment interval
Hypotension (Cardiac disorders) | 2 | 1 | 3 | 3 — Mean arterial blood pressure <65 mmHg or systolic blood pressure <100 mmHg during the 72 h treatment interval

LIMITATIONS AND CAVEATS:
Slow recruitment: switch from monocentric to 2-center study; longer than anticipated duration of the study; eventually termination of the study after only 34 of the originally intended 80 patients had been included resulting in an underpowered study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT01973335/Prot_SAP_000.pdf